CLINICAL TRIAL: NCT06457009
Title: Population Medicine Multimorbidity Intervention in Xishui on a Suspected Asthma Population: a Cluster Randomized Controlled Trial
Brief Title: Impact of Multi-Component Intervention on Suspected Asthma Population
Acronym: POPMIX-Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Simiao Chen, Professor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAMS&PUMC-IEC-2024-041
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Multimorbidity; Chronic Asthma; Population Medicine
Keywords: Suspected Asthma; Multimorbidity Interventions and Management; Clustered RCT; Pay-for-population Mechanism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Within the intervention arm, all medical practitioners will be incentivized by a pay-for-population mechanism within their township. First, finish a ECRHS questionnaire with notification of suspected asthma risk status. Those noticed will be given a face-to-face survey, simple physical examination, pulmonary function tests, and provide a multi-component intervention at baseline. For suspected asthma population, we provide community-based spirometry PFT and education; If individuals whose FEV1 improved by ≥12% and ≥200 mL, they will be undiagnosed asthma patients and encouraged to seek treatment to the superior hospitals. We provide (1) two digital health intervention programs to smokers and individuals with mental health issues; (2) CBT-based health education for study participants with abnormal BMI; (3) active recruitment into National Essential Public Health Program for those with abnormal blood pressure and glucose. Intensive follow-ups will be conducted at month 3, 6, 12.
  Interventions: Combination Product: Multi-component Intervention Package
- Control Arm (No Intervention): Those who are assigned in the control arm, we will ask them to finish the same ECRHS asthma screening online questionnaire with notification of his or her suspected asthma status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given.

INTERVENTIONS:
Combination Product: Multi-component Intervention Package — 1. Community-based spirometry pulmonary function tests and result interpretations and health education for asthma;
  2. A digital health intervention program, NicQuit, for smokers(very familiar with intelligent mobile phone);
  3. A digital health intervention program, EmoEase, for individuals whose WEMWBS questionnaire score is lower than 45(very familiar with intelligent mobile phone);
  4. Health education to smokers for smoking cessation;
  5. Health education to individuals with mental health issues;
  6. Encouragement to seek professional medication treatment in superior hospitals for undiagnosed asthma patients;
  7. To actively include individuals whose blood pressure's higher than 140/90 mmHg or/and whose random blood glucose higher than 11.1 mmol/L into the National Essential Public Health Service in China;
  8. A CBT-based health education to the BMI abnormal, i.e., BMI > 24.0 or BMI < 18.5;
  9. Pay-for-population mechanism for medical practitioners.
  Arms: Intervention arm

SUMMARY:
Study Participants: Suspected asthma population, defined as individuals whose score of asthma screening questionnaire used in ECRHS study exceeds 0 and whose age is 35 and above.

Intervention: Within the intervention arm, we have constructed a population-based pay-for-performance mechanism to encourage medical practitioners to care for population health. For study participants in the intervention arm, we will ask them to finish an online ECRHS questionnaire with notification of his or her suspected asthma status. Individuals whose score of ECRHS asthma screening exceeds 0 will be given a face-to-face survey, simple physical examination, pulmonary function tests, and provide a multi-component intervention at baseline. For suspected asthma population in the intervention arm, we provide community-based spirometry pulmonary function test (PFT) and education; If individuals whose FEV1 improved by ≥12% and ≥200 mL following bronchodilator administration with 400 ug salbutamol, they will be spirometry-defined undiagnosed asthma patient and will be encouraged to seek treatment and medication to the superior hospitals. Additionally, we provide (1) two digital health intervention programs to smokers and individuals with mental health issues; (2) CBT-based health education for study participants with abnormal BMI; (3) active recruitment into National Essential Public Health Program in China for those with abnormal blood pressure and blood glucose. Intensive follow-ups will be conducted at month 3 (telephone interview), month 6 (face-to-face with full steps of physical examination), and month 12.

Comparison: Those who are assigned in the control arm, we will ask them to finish the same ECRHS online questionnaire with notification of his or her suspected asthma status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given.

Outcomes: The primary outcomes are asthma knowledge, lung function testing, and ACT score at month 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 and above;
* Score of ECRHS asthma screening questionnaire exceeds 0;
* Residents who have lived in one township over the past 3 months and plan to reside in the same township in the upcoming year;
* Finished the informed consent

Exclusion Criteria:

* Pregnancy and other conditions that are not allowed to finish pulmonary function tests;
* Severe cognitive disorder or total loss of capability of daily living

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7400 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Chronic Diseases Controlled | 1 year
  Among all objectively measured diseases (asthma, COPD, BMI, hypertensions, type 2 diabetes, depression symptoms, anxiety symptoms), the number of chronic diseases controlled defined by objective measurement at month 12.
Lung function testing | 1 year
  Definition: Have you ever had a pulmonary function test?; Variable type: Binary; Measurement: Respondent's answer to the question;
ACT score | 1 year
  Definition: Asthma Control Test score Variable type: Continuous; Measurement: Respondent's answer to the question; Introduction to ACT score: Asthma control test (ACT), ranging from 0 to 25, the lower the score, the better asthma controlled.

SECONDARY OUTCOMES:
Self-rated health status | 1 year
  Definition: General self-assessed health status; Variable type: Continuous; Measurement: EQ-5D scale; Introduction to EQ-5D-5L scale: The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The scale could be transferred to health utility value, ranging from 0 to 1 continuously. 0 represents death and 1 represents perfect health.
Asthma Knowledge | 1 year
  Definition: The first 7 questions within Chinese version Patient Asthma Knowledge Questionnaire, the higher the score, the more correct statements the respondents will have chosen.
  Variable type: Continuous; Measurement: Respondent's answer to the question;
Bronchial Asthma Screening | 1 year
  Definition: Have you ever been screened for bronchial asthma by a doctor? Variable type: Binary; Measurement: Respondent's answer to the question;
Bronchial Asthma Diagnosis | 1 year
  Definition: Have you ever been diagnosed with bronchial asthma? Variable type: Binary; Measurement: Respondent's answer to the question;
Bronchial Asthma Treatment | 1 year
  Definition: Have you followed the treatment therapy from the professional physicians for asthma? Variable Type: Binary; Measurement: Respondent's answer to the question;
Bronchial Asthma Control | 1 year
  Definition: ACT score to categorize whether controlled or not Variable Type: Binary; Measurement: Respondent's answer to the question;
Blood pressure | 1 year
  Definition: Systolic and diastolic blood pressure (mmHg); Variable type: Continuous; Measurement: Omron portable automatic blood pressure monitor;
Blood Glucose | 1 year
  Definition: Reference standard for average plasma glucose concentration over a period of time; Variable type: Continuous; Measurement: Blood glucose meter;
Waist circumference | 1 year
  Definition: Waist circumference (cm); Variable type: Continuous; Measurement: Soft measuring tape;
BMI | 1 year
  Definition: Body mass index (BMI), weight divided by height squared (kg/m²); Variable type: Continuous; Measurement: Calculation;
Number of Outpatient Visits | 1 year
  Definition: Outpatient visits and type of hospital; Variable type: Count; Measurement: Survey data/insurance/outpatient data;
Number of Inpatient Visits | 1 year
  Definition: Inpatient visits and type of hospital; Variable type: Count; Measurement: Survey data/insurance/outpatient data;
Medical expenditure within a family over the past year | 1 year
  Definition: Healthcare-related expenditures; Variable type: Continuous; Measurement: Survey data/insurance/outpatient/inpatient data;
Depression Symptoms | 1 year
  Definition: Emotional disorders, including sadness, loss, and anger; Variable type: Continuous; Measurement: PHQ-9; Introduction to PHQ-9: Patient Health Questionnaire- 9 items (PHQ-9), ranging from 0 to 27, the higher the score, the severer the depression symptoms for the respondents will be.
Anxiety Symptoms | 1 year
  Definition: Unpleasant state of inner turmoil; Variable type: Continuous; Measurement: GAD-7; Introduction to GAD-7: General Anxiety Disorder - 7 (GAD-7), ranging from 0 to 21, the higher the score, the severer the anxiety symptoms for the respondents will be.
Warwick-Edinburgh Mental Well-being Scale, WEM -WBS score | 1 year
  Definition: Reflects overall mental health problems; Variable type: Continuous; Measurement: WEMWBS; Introduction to WEMWBS: Warwick-Edinburgh Mental Well-being Scale, ranging from 14 to 70, the lower the score, the worse one's general mental health will be.
Family level annual consumption expenditure | 1 year
  Definition: Annual total household expenditure Variable type: Categorical Measurement: Answer to a question covering local expenditure categories by the household representative
Employment status | 1 year
  Definition: Main occupation and type; Variable type: Categorical; Measurement: Respondent's answer to the question;
Productivity Loss | 1 year
  Definition: Productivity loss due to illness or health problems from Working Productivity and Activity Impairment-General Health Chinese version 2.0; Variable type: Continuous; Measurement: Respondent's answer to the question;
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Questions:
  1. = currently employed
  2. = hours missed due to health problems
  3. = hours missed other reasons
  4. = hours actually worked
  5. = degree health affected productivity while working
  6. = degree health affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages.
  Percent work time missed due to health: Q2/(Q2+Q4)
  Percent impairment while working due to health: Q5/10
  Percent overall work impairment due to health:
  Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]
  Percent activity impairment due to health: Q6/10
FEV1 measurement | 1 year
  Definition: Forced Expiratory Volume in one second (FEV1); Variable type: Continuous; Measurement: Pulmonary function test, portable spirometry;
HBP Screening | 1 year
  Definition: Have you ever had your blood pressure measured by a doctor, nurse, or other healthcare professional? Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Diagnosis | 1 year
  Definition: Have you ever been diagnosed with hypertension by a doctor? Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Treatment | 1 year
  Definition: Are you currently taking any antihypertensive medication prescribed by a doctor or other healthcare professional? Variable type: Binary Measurement: Respondent's answer to the question
HBP Control | 1 year
  Definition: Blood pressure within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood pressure measurement;
T2DM Screening | 1 year
  Definition: Have you ever had your blood glucose measured by a doctor, nurse, or other healthcare professional? Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Diagnosis | 1 year
  Definition: Have you ever been diagnosed with T2DM by a doctor? Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Treatment | 1 year
  Definition: Are you currently receiving a type 2 diabetes treatment plan prescribed by a doctor or other healthcare professional? Variable type: Binary Measurement: Respondent's answer to the question
T2DM Control | 1 year
  Definition: Blood glucose within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood glucose measurement;
Smoking Status | 1 year
  Definition: Do you currently smoke? Variable type: Binary; Measurement: Respondent's answer to the question
  ;
Smoking Amount | 1 year
  Definition: How many cigarettes do you smoke per day on average? Variable type: Count; Measurement: Respondent's answer to the question;
Drinking Status | 1 year
  Definition: Frequency of alcohol consumption in the past 3 months; Variable type: Categorical; Measurement: Respondent's answer to the question;
Sugar Consumption | 1 year
  Definition: Frequency of consumption of sugary foods/drinks; Variable type: Categorical; Measurement: Respondent's answer to the question;
Salted Vegetables Consumption | 1 year
  Definition: Frequency of consumption of salty vegetables; Variable type: Categorical; Measurement: Respondent's answer to the question;
Vegetable Consumption | 1 year
  Definition: Frequency of consumption of vegetable; Variable type: Categorical; Measurement: Respondent's answer to the question;
Physical exercise | 1 year
  Definition: Hours of physical exercise per week; Variable type: Count; Measurement: Respondent's answer to the question;
Self-awareness of COPD | 1 year
  Definition: Have you ever been diagnosed with COPD? Variable type: Binary; Measurement: Respondent's answer to the question;
COPD-Knowledge | 1 year
  Definition: COPD Knowledge Questionnaire(Excerpt); Variable type: Continuous; Measurement: Respondent's answer to the questions;
mMRC score | 1 year
  Definition: score for mMRC questionnaire Variable type: Categorical Measurement: Respondent's answers to the question Introduction to mMRC: Modified Medical Research Council, categorical value, level 0 represents a good respiratory condition, while the maximum level 4 represents a very bad respiratory condition.
Smoking Dependence | 1 year
  Fagerström test for nicotine dependence (FTND) is a scale that measures the nicotine dependence of smokers, ranging from 0 to 15, the higher the value, the worse the nicotine dependence will be. Heaviness Index of Smoking (HIS) could also be calculated using part of the scale, ranging from 0 to 6, and higher score means worse nicotine dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Simiao Chen, Ph.D., Principal Investigator — Peking Union Medical College
Locations (1):
- Xishui County for Xishui Trial, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No